CLINICAL TRIAL: NCT01277601
Title: A Phase 4, Randomized, Open-label, Active-Controlled, Superiority Study to Evaluate the Efficacy and Safety of Tenofovir Disoproxil Fumarate (TDF) in Combination With Peginterferon α-2a (Pegasys®) Versus Standard of Care Tenofovir Disoproxil Fumarate Monotherapy or Peginterferon α-2a Monotherapy for 48 Weeks in Non-Cirrhotic Subjects With HBeAg-Positive or HBeAg-Negative Chronic Hepatitis B (CHB)
Brief Title: Efficacy & Safety of Tenofovir Disoproxil Fumarate (TDF) Plus Peginterferon α-2a (Peg-IFN) Versus TDF or Peg-IFN Monotherapy in Chronic Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-174-0149; 2010-024586-45 (EudraCT Number)
Record Dates: First submitted 2011-01-13; First posted 2011-01-17 (Estimated); Results first posted 2015-09-09 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic Hepatitis B; Hep B; Non cirrhotic; Tenofovir disoproxil fumarate (TDF); Peginterferon α-2a (Peg-IFN)
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- TDF+Peg-IFN 48 Weeks (Experimental): TDF plus Peg-IFN for 48 weeks
  Interventions: Drug: TDF; Drug: Peg-IFN
- TDF 48 Weeks + Peg-IFN 16 Weeks (Experimental): TDF plus Peg-IFN for 16 weeks, followed by TDF alone for an additional 32 weeks
  Interventions: Drug: TDF; Drug: Peg-IFN
- TDF 120 Weeks (Active Comparator): TDF monotherapy for 120 weeks
  Interventions: Drug: TDF
- Peg-IFN 48 Weeks (Active Comparator): Peg-IFN monotherapy for 48 weeks
  Interventions: Drug: Peg-IFN

INTERVENTIONS:
Drug: TDF — TDF 300 mg tablets administered orally once daily
  Other Names: Viread®
  Arms: TDF 120 Weeks; TDF 48 Weeks + Peg-IFN 16 Weeks; TDF+Peg-IFN 48 Weeks
Drug: Peg-IFN — Peg-IFN 180 µg administered via subcutaneous injection once weekly
  Other Names: Pegasys®
  Arms: Peg-IFN 48 Weeks; TDF 48 Weeks + Peg-IFN 16 Weeks; TDF+Peg-IFN 48 Weeks

SUMMARY:
The primary objective of this study is to evaluate the efficacy of tenofovir disoproxil fumarate (TDF) plus peginterferon α-2a (Peg-IFN) combination therapy for 48 weeks versus standard of care TDF monotherapy or Peg-IFN monotherapy for 48 weeks in non-cirrhotic adults with chronic hepatitis B virus (HBV) as determined by loss of hepatitis B surface antigen (HBsAg).

The study will consist of 2 phases for participants in the TDF+Peg-IFN 48 Weeks, TDF 48 Weeks + Peg-IFN 16 Weeks, and Peg-IFN 48 Weeks groups. Following an initial 48 weeks of treatment, participants in these groups will be monitored for 24 weeks for signs of worsening HBV, and those meeting TDF retreatment and flare management criteria will be eligible to receive TDF monotherapy during a retreatment phase, up to Week 120.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18-75) with chronic HBV (positive for serum hepatitis B surface antigen (HBsAg) or HBV DNA for at least 6 months) prior to baseline
* Anti-HBV treatment-naive adults; adults who have taken oral anti-HBV nucleoside therapy with the last dose ≥ 24 weeks prior to screening are also eligible.
* Positive or negative for hepatitis B e antigen (HBeAg)
* HBV DNA ≥ 20,000 IU/ml (HBeAg-positive participants) and ≥ 2,000 IU/ml (HBeAg-negative participants)
* Alanine aminotransferase (ALT) > 54 U/L and ≤ 400 U/L for men and > 36 U/L and ≤ 300 U/L for women
* Creatinine clearance ≥ 70 mL/min
* Negative serum pregnancy test for females of childbearing potential
* Sexually active females of childbearing potential must agree to use a protocol-recommended method of contraception throughout the study and for 30 days following the last dose of study medication
* Lactating females must agree to discontinue nursing before initiation of study investigational medicinal product

Exclusion Criteria:

* Known bridging fibrosis or cirrhosis and/or decompensated liver disease
* Evidence of hepatocellular carcinoma
* Significant kidney, heart, lung, neurological, autoimmune disease, or bone disease (eg, osteomalacia,chronic osteomyelitis, osteogenesis imperfecta, osteochondrosis, multiple bone fractures)
* Absolute neutrophil count < 1,500/mm^3, platelet < 100,000/mm^3, hemoglobin < 10 g/dL (female) or < 11 g/dL (male)
* History of severe depression or severe psychiatric disease
* Thyroid dysfunction
* Coinfection with HIV, hepatitis C virus (HCV) or hepatitis D virus (HDV)
* Pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 751 (Actual)
Dates: Start 2011-04; Primary Completion 2014-08 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Jump, Study Director — Gilead Sciences
Locations (171):
- United States (26):
  - Asian Pacific Liver Center, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - Research and Education Inc, San Diego, California
  - San Jose Gastroenterology, San Jose, California
  - Avail Clinical Research, LLC, DeLand, Florida
  - Centre for Advanced Gastroenterology, Maitland, Florida
  - University of Miami / Jackson Memorial Medical Center, Miami, Florida
  - University of Chicago, Chicago, Illinois
  - LSU Gastroenterology/Center for Digestive Diseases, New Orleans, Louisiana
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Digestive Disease Associates, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - ID Care, Inc., Hillsborough, New Jersey
  - Medical Procare, PLLC, Flushing, New York
  - North Shore University Hospital, Great Neck, New York
  - Beth Israel Medical Center, New York, New York
  - New York Univ. Medical Center, New York, New York
  - Weill Cornell Medical College of Cornell University, New York, New York
  - Private Practice, Philadelphia, Pennsylvania
  - Advanced Liver Therapies at St. Luke's Episcopal Hospital, Houston, Texas
  - Kelsey Research Foundation, Houston, Texas
  - Liver Associates of Texas,, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Liver Institute of Virginia, Bon Secours Health System, Richmond, Virginia
  - McGuire Research Institute, Richmond, Virginia
- Australia (19):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Saint George's Hospital, Kogarah, New South Wales
  - Liverpool Hospital,Gastroenterology Department, Liverpool, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Center, Adelaide, South Australia
  - Royal Adelaide Hospital, Adelaide SA, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Saint Vincents Hospital, Fitzroy, Victoria
  - Western Hospital, Footscray, Victoria
  - Austin Health, Heidelberg, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Box Hill Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Fremantle Hospital, Fremantle
  - Sir Charles Gairdner Hospital, Nedlands
  - Royal Perth Hospital, Perth
- Canada (8):
  - Heritage Med Research Clinic, Univ of Calgary, Calgary, Alberta
  - University of Alberta, Zeidler Ledcore Centre, Zeidler Ledcore Centre, Alberta
  - Gastrointestional Research Institute, Vancouver, British Columbia
  - Gordon & Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - Liver and Intestinal Research Centre, Vancouver, British Columbia
  - The Ottawa Hospital,Division of Infectious Diseases, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Liver Centre, Toronto, Ontario
- France (8):
  - Hôpital Beaujon, Service Hepatologie- Centre Pierre Abrami, Clichy, Cedex
  - Hôpital de la Croix Rousse, Lyon, Cedex
  - Hopital Tenon, Paris
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - Hopital Charles Nicolle, Rouen
  - Centre Hospitalier Regional et Universitaire de Strasbourg, Hopital Civil, Strasbourg
  - Centre Hospitalier Universitaire Purpan, Toulouse
  - Hopital Paul Brousse, Villejuif
- Germany (8):
  - Johannes Gutenberg-Universitat Mainz,, Mainz, Rhineland-Palatinate
  - Charite Berlin, Berlin
  - Universitatsklinik Koln, Cologne
  - Universitätsklinikum Essen - klinikum für Gastroenterolgie und Hepatologie,, Essen
  - Johann-Wolfgang-Goethe Universitat,, Frankfurt
  - Asklepios Westklinikum, Hamburg
  - Medizinische Hochschule Hannover,Hastroenterologie und Hepatologie, Hanover
  - Universitatsklinikum Leipzig, Leipzig
- Greece (4):
  - Ippokratio Hospital Salonica, Thessaloniki, Attica
  - Ippokratio Hospital Athens, Attica
  - General University Hospital of Patras, Pátrai
  - Hippokration General Hospital of Thessaloniki, Thessaloniki
- Hong Kong (4):
  - Queen Mary Hospital, Hong Kong
  - Princess Margaret Hospital, Kowloon
  - Prince of Wales Hospital, Shatin
  - Alice Ho Miu Ling Nethersole Hospital, Tai Po
- India (13):
  - Global Hospital, Lakdi Ka Pul, Hyderabad, Andhra Pradesh
  - Institute of digestive and liver disease, Dispur Hospital Ganeshguri, Guwahati, Assam
  - Vedanta Institute of Medical Sciences, Ahmedabad, Gujarat
  - Liver Clinic, Surat, Gujarat
  - Manipal Hospitals, Bangalore, Karnataka
  - Department of Hepatology, Institute of Liver Diseases, HPB Surgery and Transplant, Global Hospital, Mumbai, Maharashtra
  - Seth GS Medical College and KEM Hospital, Acharya Donde Marg,Parel, Mumbai, Maharashtra
  - Midas Institute of Gastroenterology, Nagpur, Maharashtra
  - Dharamasi Hospital,Chandni Chowk, South Shivajinagar,, Sangli, Maharashtra
  - All India Institute of Medical Sciences, Ansari Nagar, Delhi, New Delhi
  - Institute of Liver and Biliary Sciences, New Delhi, New Delhi
  - VGM Hospital, Coimbatore, Tamil Nadu
  - Institute of Post Graduate Medical Education And Research, Kolkata, West Bengal
- Italy (8):
  - Azienda Ospedaliero-Universitaria di Cagliari, Monserrato, Cagliari
  - Fondazione IRCCS Ca Granda - Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele, Milan
  - Seconda Universita degli Studi di Napoli, Napoli
  - Azienda Ospedaliera di Parma,Department of Infectious Diseases and hepatology, Parma
  - Fondazione PTV - Policlinico Tor Vergata, Roma
  - Policlinico Umberto I, Rome
  - University of Milan,Azienda Ospedaliera San Giovanni, Battista di Torino,Dipartimento di Gastroenterologia, Torino
- Netherlands (3):
  - Academisch Medisch Centrum, Amsterdam
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Erasmus Medisch Centrum, Rotterdam
- Poland (8):
  - Samodzielny Publiczny Szpital Kliniczny 1,Klinika Chorób Zakaznych,ulica Staszica 16, Lublin, Lublin Voivodeship
  - Szpital Specjalistyczny w Chorzowie, Chorzów, Silesian Voivodeship
  - Wojewodzki Szpital Specjalistyczny Kazimierza Dluskeigo w Bialymstoku, Bialystok
  - Wojewódzki Szpital Obserwacyjno Zakazny im. Tadeusza Browicza, Bydgoszcz
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Wojewódzki Specjalistyczny Szpital im. Dr Wladyslawa Bieganskiego w Lodzi, Lodz
  - SP ZOZ Wojewodzki Szpital Zakazny, Warsaw
  - Wojewódzki Specjalistyczny Szpital im. Dr Wladyslawa Bieganskiego w Lodzi, Lodz, Łódź Voivodeship
- Portugal (4):
  - Hospital de Egas Moniz, Lisbon
  - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar do Porto, Porto
  - Hospital São João, Porto
- Romania (7):
  - Neomed Research, Brasov
  - Institutul National de Boli Infectioase "Prof. Dr. Matei Bals", Bucharest
  - Institutul National de Boli Infectioase Prof.Dr. Matei Bals, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Spitalul Clinic de Boli Infectioase si Tropicale "Dr. Victor Babes", Bucharest
  - Spitalul Clinic Judetean de Urgenta Sibiu, Sibiu
  - Cabinet Particular Policlinic Algomed SRL-Gastroenterologie, Timișoara
- Singapore (4):
  - Changi General Hospital, Singapore
  - National University Hospital Singapore, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (18):
  - SoonChunHyang University Hospital Cheonan, Cheonan, Chungcheon
  - Yonsei Unversity Wonju College of Medicine Wonju Christian Hospital, Wŏnju, Gangwon-do
  - Korea University Ansan Hospital, Ansan-si, Gyeonggi-d
  - Bucheon St. Mary's Hospital, Bucheon-si, Gyeonggi-d
  - Korea University Guro Hospital, Seoul, Gyeonggi-d
  - CHA Bundang Medical Center, CHA University, Sungnam, Gyeonggi-d
  - Pusan National University Hospital, Busan, Gyeongsang
  - Kyungpook National University Hospital, Daegu, Gyeongsang
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsang
  - Inje University Busan Paik Hospital, Busan
  - Inje University Ilsan Paik Hospital, Goyang, Gyeonggi-Do
  - Digestive Disease Cntr, Konkuk Univ Hosp, Kwangjin-gu, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul Saint Mary's Hospital, Seoul
- Spain (6):
  - Hospital Universitario de La Princesa, Madrid, Madrid
  - Hospital General Universitari Vall d' Hebron, Barcelona
  - Hospital Carlos III, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Meixoeiro, Vigo, Pontevedra
- Taiwan (14):
  - Far-Eastern Memorial Hosp, New Taipei City, Banciao Dist
  - Chang Gung Medical Foundation.LinKou Branch, Taoyuan District, Taoyuan
  - Changhua Christain Hospital, Changhua
  - Chiayi Christian Hosp, Chiayi City
  - Buddhist Tzu Chi General Hospital, Hualien City
  - Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University Hospital, Kaosiung
  - Chang Gung Medical Foundation-Keelung, Keelung Town/KEELUNG CITY
  - China Medical University Hospital, Taichung
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans Genl Hosp, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Cathay General Hospital, Taipei
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (5):
  - Ankara Üniversitesi Tip Fakültesi, Ankara, Ankara
  - Hacettepe Üniversitesi Tip Fakültesi, Ankara, Ankara
  - Gaziantep Üniversitesi Tip Fakültesi, Sahinbey Arastirma ve Uygulama Hastanesi, Gaziantep
  - Istanbul Universitesi Istanbul Tip Fakultesi, Istanbul
  - Mersin Üniversitesi Tip Fakültesi, Saglik Arastirma ve Uygulama Hastanesi, Mersin
- United Kingdom (4):
  - The Queen Elizabeth Hospital, Birmingham, Wstmid
  - Royal Free Hospital, Hampstead,London
  - Barts and The London NHS Trust, London
  - King's College Hospital, London

REFERENCES:
- [Result] Marcellin P, Ahn SH, Ma X, Caruntu FA, Tak WY, Elkashab M, Chuang WL, Lim SG, Tabak F, Mehta R, Petersen J, Foster GR, Lou L, Martins EB, Dinh P, Lin L, Corsa A, Charuworn P, Subramanian GM, Reiser H, Reesink HW, Fung S, Strasser SI, Trinh H, Buti M, Gaeta GB, Hui AJ, Papatheodoridis G, Flisiak R, Chan HL; Study 149 Investigators. Combination of Tenofovir Disoproxil Fumarate and Peginterferon alpha-2a Increases Loss of Hepatitis B Surface Antigen in Patients With Chronic Hepatitis B. Gastroenterology. 2016 Jan;150(1):134-144.e10. doi: 10.1053/j.gastro.2015.09.043. Epub 2015 Oct 8. PMID 26453773
- [Result] Chan HL, Elkhashab M, Trinh H, Tak WY, Ma X, Chuang WL, Kim YJ, Martins EB, Lin L, Dinh P, Charuworn P, Foster GR, Marcellin P. Association of baseline vitamin D levels with clinical parameters and treatment outcomes in chronic hepatitis B. J Hepatol. 2015 Nov;63(5):1086-92. doi: 10.1016/j.jhep.2015.06.025. Epub 2015 Jul 2. PMID 26143444

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Europe, Asia, and Australia. The first participant was screened on 12 April 2011. The last study visit occurred on 17 July 2015.
Pre-assignment Details: 1597 participants were screened.
Groups:
- TDF+Peg-IFN 48 Weeks: Tenofovir disoproxil fumarate (TDF) 300 mg tablet once daily plus peginterferon α-2a (Peg-IFN) 180 µg subcutaneous (s.c.) injection once weekly for 48 weeks
- TDF 48 Weeks + Peg-IFN 16 Weeks: TDF 300 mg tablet once daily plus Peg-IFN 180 µg s.c. injection once weekly for 16 weeks followed by TDF 300 mg tablet once daily for an additional 32 weeks
- TDF 120 Weeks: TDF 300 mg tablet once daily for 120 weeks
- Peg-IFN 48 Weeks: Peg-IFN 180 µg s.c. injection once weekly for 48 weeks
Period: Overall Study
Arm/Group | TDF+Peg-IFN 48 Weeks | TDF 48 Weeks + Peg-IFN 16 Weeks | TDF 120 Weeks | Peg-IFN 48 Weeks
Started | 188 | 187 | 190 | 186
Completed | 151 | 139 | 163 | 150
Not Completed | 37 | 48 | 27 | 36
Not completed — Adverse Event | 5 | 3 | 0 | 7
Not completed — Withdrawal by Subject | 18 | 21 | 8 | 17
Not completed — Lost to Follow-up | 7 | 9 | 4 | 2
Not completed — Physician Decision | 3 | 5 | 1 | 6
Not completed — Pregnancy | 2 | 2 | 4 | 1
Not completed — Noncompliance with Study Drug | 1 | 3 | 2 | 0
Not completed — Subject Never Dosed with Study Drug | 1 | 2 | 3 | 1
Not completed — Protocol Violation | 0 | 2 | 5 | 0
Not completed — Subject Terminated from Study by Sponsor | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized and received at least 1 dose of study drug. Participants were analyzed by actual treatment received.
  11 participants were never dosed are not included in the Safety Analysis Set due to the following reasons for discontinuation: 7 = Subject Never Dosed with Study Drug; 4 = Withdrawal by Subject.
Groups:
- TDF+Peg-IFN 48 Weeks: TDF 300 mg tablet once daily plus Peg-IFN 180 µg s.c. injection once weekly for 48 weeks
- TDF 48 Weeks + Peg-IFN 16 Week: TDF 300 mg tablet once daily plus Peg-IFN 180 µg s.c. injection once weekly for 16 weeks followed by TDF 300 mg tablet once daily for an additional 32 weeks
- Total: Total of all reporting groups
Arm/Group | TDF+Peg-IFN 48 Weeks | TDF 48 Weeks + Peg-IFN 16 Week | TDF 120 Weeks | Peg-IFN 48 Weeks | Total
Number analyzed (Participants) | 186 | 184 | 185 | 185 | 740
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (10.7) | 37 (9.9) | 36 (10.8) | 38 (10.5) | 37 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 65 | 64 | 66 | 254
  Male | 127 | 119 | 121 | 119 | 486
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 3 | 7 | 18
  Not Hispanic or Latino | 182 | 179 | 181 | 177 | 719
  Unknown or Not Reported | 0 | 1 | 1 | 1 | 3
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 142 | 134 | 141 | 137 | 554
  Black or African American | 5 | 3 | 4 | 6 | 18
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 1 | 3
  White | 36 | 45 | 39 | 41 | 161
  Other | 1 | 2 | 1 | 0 | 4
Region of Enrollment [Number; unit: participants]
  Romania | 12 | 15 | 13 | 9 | 49
  Singapore | 7 | 5 | 7 | 8 | 27
  Hong Kong | 25 | 24 | 27 | 21 | 97
  United States | 19 | 17 | 23 | 26 | 85
  United Kingdom | 2 | 3 | 1 | 4 | 10
  Portugal | 0 | 3 | 0 | 0 | 3
  India | 10 | 5 | 9 | 6 | 30
  Spain | 3 | 3 | 3 | 5 | 14
  Greece | 0 | 3 | 2 | 4 | 9
  Canada | 19 | 14 | 14 | 11 | 58
  Netherlands | 2 | 1 | 0 | 1 | 4
  Turkey | 5 | 6 | 6 | 7 | 24
  Taiwan | 20 | 15 | 12 | 19 | 66
  Korea, Republic of | 34 | 38 | 38 | 35 | 145
  Poland | 4 | 7 | 6 | 5 | 22
  Italy | 2 | 1 | 4 | 4 | 11
  Australia | 10 | 14 | 15 | 14 | 53
  France | 6 | 3 | 1 | 3 | 13
  Germany | 6 | 7 | 4 | 3 | 20
Hepatitis B Surface Antigen (HBsAg) [Mean (Standard Deviation); unit: log 10 IU/mL] | 3.88 (0.840) | 3.84 (0.849) | 3.89 (0.812) | 3.76 (0.844) | 3.84 (0.836)
Hepatitis B e Antigen (HBeAg) Status [Number; unit: participants]
  Reactive | 108 | 105 | 109 | 106 | 428
  Nonreactive | 78 | 79 | 76 | 79 | 312
Hepatitis B Virus (HBV) DNA [Mean (Standard Deviation); unit: log 10 IU/mL] | 7.06 (1.542) | 7.13 (1.505) | 7.02 (1.550) | 6.94 (1.619) | 7.04 (1.553)
HBV Genotype [Number; unit: participants]
  Genotype A | 17 | 16 | 14 | 14 | 61
  Genotype B | 50 | 51 | 49 | 53 | 203
  Genotype C | 78 | 79 | 78 | 79 | 314
  Genotype D | 39 | 36 | 41 | 38 | 154
  Genotype E-H | 2 | 2 | 3 | 1 | 8
Alanine Aminotransferase (ALT) [Mean (Standard Deviation); unit: U/L] | 121.2 (180.82) | 112.2 (94.44) | 100.9 (67.65) | 106.6 (91.51) | 110.3 (116.94)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HBsAg Loss at Week 72 Following Treatment With 48 Weeks of TDF Plus Peg-IFN Combination Versus Peg-IFN Alone for 48 Weeks or TDF Alone
Description: Loss of HBsAg was defined as change of detectable HBsAg from positive to negative. Proportions are based on a Kaplan-Meier estimate.
  The analysis visit window for Week 72 comprised Week 70 through Week 78, so results up to Week 78 are included in this analysis.
Time Frame: Baseline; Week 72
Population: Full Analysis Set: participants who were randomized and received at least 1 dose of study drug. Participants in the TDF+Peg-IFN 48 Weeks, TDF 120 Weeks, and Peg-IFN 48 Weeks groups were analyzed by randomized treatment.
Measure: Number; unit: percentage of participants
Arm/Group | TDF+Peg-IFN 48 Weeks | TDF 120 Weeks | Peg-IFN 48 Weeks
Number analyzed (Participants) | 186 | 185 | 185
percentage of participants | 9.05 | 0.00 | 2.84
Statistical Analysis 1: Comparison: TDF+Peg-IFN 48 Weeks vs TDF 120 Weeks; Test type: Superiority or Other; p < 0.001, Log Rank — Raw p-values comparing treatments were based on a log-rank test stratified by HBeAg status and viral genotype
Statistical Analysis 2: Comparison: TDF+Peg-IFN 48 Weeks vs Peg-IFN 48 Weeks; Test type: Superiority or Other; p = 0.002, Log Rank — Raw p-values comparing treatments were based on a log-rank test stratified by HBeAg status and viral genotype

2. Secondary Outcome: Percentage of Participants With HBsAg Loss at Week 72 Following Treatment With TDF (48 Weeks) Plus Peg-IFN (16 Weeks) Combination Versus Peg-IFN Alone for 48 Weeks or TDF Alone
Description: as for outcome 1
Time Frame: Baseline; Week 72
Population: Full Analysis Set. Participants in the TDF 48 week + Peg-IFN 16 Weeks, TDF 120 Weeks, and Peg-IFN 48 Weeks groups were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TDF 48 Weeks + Peg-IFN 16 Weeks | TDF 120 Weeks | Peg-IFN 48 Weeks
Number analyzed (Participants) | 184 | 185 | 185
percentage of participants | 2.83 | 0.00 | 2.84

3. Secondary Outcome: Percentage of Participants With HBsAg Loss at Weeks 96 and 120
Description: Loss of HBsAg was defined as change of detectable HBsAg from positive to negative. Proportions are based on a Kaplan-Meier estimate.
  The analysis visit window for Week 96 comprised study Week 90 through Week 102, so results up to Week 102 are included in this analysis. The analysis visit window for Week 120 comprised study Week 114 through Week 126, so results up to Week 126 are included in this analysis.
Time Frame: Baseline; Weeks 96 and 120
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Groups:
- TDF 120 Week: TDF 300 mg tablet once daily for 120 weeks
Arm/Group | TDF+Peg-IFN 48 Weeks | TDF 48 Weeks + Peg-IFN 16 Weeks | TDF 120 Week | Peg-IFN 48 Weeks
Number analyzed (Participants) | 186 | 184 | 185 | 185
percentage of participants
  Week 96 | 9.69 | 3.49 | 0.00 | 2.84
  Week 120 | 10.36 | 3.49 | 0.00 | 3.51

4. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion at Weeks 72, 96, and 120
Description: HBsAg seroconversion was defined as change of detectable antibody to HBsAg from negative to positive. Proportions are based on a Kaplan-Meier estimate.
  The analysis visit window for Week 72 comprised Week 70 through Week 78, so results up to Week 78 are included in this analysis. The analysis visit window for Week 96 comprised Week 90 through Week 102, so results up to Week 102 are included in this analysis. The analysis visit window for Week 120 comprised Week 114 through Week 120.
Time Frame: Baseline; Weeks 72, 96, and 120
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | TDF+Peg-IFN 48 Weeks | TDF 48 Weeks + Peg-IFN 16 Weeks | TDF 120 Weeks | Peg-IFN 48 Weeks
Number analyzed (Participants) | 186 | 184 | 185 | 185
percentage of participants
  Week 72 | 8.05 | 0.56 | 0.00 | 2.87
  Week 96 | 8.05 | 0.56 | 0.00 | 2.87
  Week 120 | 10.08 | 0.56 | 0.00 | 2.87

5. Secondary Outcome: Percentage of Participants With HBeAg Loss and Seroconversion at Week 72
Description: Loss of HBeAg was defined as change of detectable HBeAg from positive to negative. HBeAg seroconversion was defined as change of detectable antibody to HBeAg from negative to positive. Percentages were based on the number of subjects with non-missing HBeAg results or missing HBeAg results imputed as failures at each visit.
  For the TDF+Peg-IFN 48 Weeks, TDF 48 Weeks + Peg-IFN 16 Weeks, and Peg-IFN 48 Weeks groups, data are presented in the "Not Retreated" column for participants who had not entered the retreatment phase by Week 72, and in the "Retreated" column for participants who did enter the retreatment phase by Week 72.
Time Frame: Baseline; Week 72
Population: Participants in the Full Analysis Set who were HBeAg reactive or indeterminate at baseline were analyzed. The missing = failure method was used in which participants on study with missing data were considered to have failed to achieve the outcome.
Measure: Number; unit: percentage of participants
Groups:
- TDF+Peg-IFN 48 Week (Not Retreated): TDF 300 mg tablet once daily plus Peg-IFN 180 µg s.c. injection once weekly for 48 weeks in the initial treatment phase
- TDF+Peg-IFN 48 Weeks (Retreated); TDF 48 Weeks + Peg-IFN 16 Weeks (Retreated); Peg-IFN 48 Weeks (Retreated): Following the randomized treatment, participants who met protocol-specified criteria were retreated with TDF 300 mg tablet once daily up to Week 120 in the retreatment phase.
- TDF 48 Weeks + Peg-IFN 16 Week (Not Retreated): TDF 300 mg tablet once daily plus Peg-IFN 180 µg s.c. injection once weekly for 16 weeks followed by TDF 300 mg tablet once daily for an additional 32 weeks in the initial treatment phase
- TDF 120 Weeks: TDF 300 mg tablet once daily for 120 weeks. Participants in this group were not eligible to enter the retreatment phase.
- Peg-IFN 48 Weeks (Not Retreated): Peg-IFN 180 µg s.c. injection once weekly for 48 weeks in the initial treatment phase
Arm/Group | TDF+Peg-IFN 48 Week (Not Retreated) | TDF+Peg-IFN 48 Weeks (Retreated) | TDF 48 Weeks + Peg-IFN 16 Week (Not Retreated) | TDF 48 Weeks + Peg-IFN 16 Weeks (Retreated) | TDF 120 Weeks | Peg-IFN 48 Weeks (Not Retreated) | Peg-IFN 48 Weeks (Retreated)
Number analyzed (Participants) | 76 | 32 | 61 | 44 | 109 | 64 | 42
percentage of participants
  HBeAg Loss | 35.5 | 15.6 | 32.8 | 15.9 | 14.7 | 32.8 | 14.3
  HBeAg Seroconversion | 28.9 | 15.6 | 31.1 | 13.6 | 12.8 | 31.3 | 14.3

6. Secondary Outcome: Percentage of Participants With HBeAg Loss and Seroconversion at Week 96
Description: Loss of HBeAg was defined as change of detectable HBeAg from positive to negative. HBeAg seroconversion was defined as change of detectable antibody to HBeAg from negative to positive. Percentages were based on the number of subjects with non-missing HBeAg results or missing HBeAg results imputed as failures at each visit.
  For the TDF+Peg-IFN 48 Weeks, TDF 48 Weeks + Peg-IFN 16 Weeks, and Peg-IFN 48 Weeks groups, data are presented in the "Not Retreated" column for participants who had not entered the retreatment phase by Week 96, and in the "Retreated" column for participants who did enter the retreatment phase by Week 96.
Time Frame: Baseline; Week 96
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | TDF+Peg-IFN 48 Week (Not Retreated) | TDF+Peg-IFN 48 Weeks (Retreated) | TDF 48 Weeks + Peg-IFN 16 Week (Not Retreated) | TDF 48 Weeks + Peg-IFN 16 Weeks (Retreated) | TDF 120 Weeks | Peg-IFN 48 Weeks (Not Retreated) | Peg-IFN 48 Weeks (Retreated)
Number analyzed (Participants) | 44 | 64 | 44 | 61 | 109 | 37 | 69
percentage of participants
  HBeAg Loss | 43.2 | 20.3 | 45.5 | 14.8 | 18.3 | 37.8 | 14.5
  HBeAg Seroconversion | 36.4 | 18.8 | 43.2 | 13.1 | 16.5 | 29.7 | 13.0

7. Secondary Outcome: Percentage of Participants With HBeAg Loss and Seroconversion at Week 120
Description: Loss of HBeAg was defined as change of detectable HBeAg from positive to negative. HBeAg seroconversion was defined as change of detectable antibody to HBeAg from negative to positive. Percentages were based on the number of subjects with non-missing HBeAg results or missing HBeAg results imputed as failures at each visit.
  For the TDF+Peg-IFN 48 Weeks, TDF 48 Weeks + Peg-IFN 16 Weeks, and Peg-IFN 48 Weeks groups, data are presented in the "Not Retreated" column for participants who had not entered the retreatment phase by Week 120, and in the "Retreated" column for participants who did enter the retreatment phase by Week 120.
Time Frame: Baseline; Week 120
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | TDF+Peg-IFN 48 Week (Not Retreated) | TDF+Peg-IFN 48 Weeks (Retreated) | TDF 48 Weeks + Peg-IFN 16 Week (Not Retreated) | TDF 48 Weeks + Peg-IFN 16 Weeks (Retreated) | TDF 120 Weeks | Peg-IFN 48 Weeks (Not Retreated) | Peg-IFN 48 Weeks (Retreated)
Number analyzed (Participants) | 44 | 64 | 40 | 65 | 109 | 36 | 70
percentage of participants
  HBeAg Loss | 38.6 | 25.0 | 37.5 | 23.1 | 20.2 | 33.3 | 18.6
  HBeAg Seroconversion | 29.5 | 21.9 | 35.0 | 15.4 | 15.6 | 25.0 | 17.1

8. Secondary Outcome: Percentage of Participants With Virological Response (HBV DNA < 117 IU/mL) at Week 72
Description: For the TDF+Peg-IFN 48 Weeks, TDF 48 Weeks + Peg-IFN 16 Weeks, and Peg-IFN 48 Weeks groups, data are presented in the "Not Retreated" column for participants who had not entered the retreatment phase by Week 72, and in the "Retreated" column for participants who did enter the retreatment phase by Week 72.
Time Frame: Week 72
Population: Full Analysis Set. The missing = failure method was used in which participants on study with missing data were considered to have failed to achieve the endpoint.
Measure: Number; unit: percentage of participants
Groups:
- TDF+Peg-IFN 48 Weeks (Not Retreated): TDF 300 mg tablet once daily plus Peg-IFN 180 µg s.c. injection once weekly for 48 weeks in the initial treatment phase
- TDF 48 Weeks + Peg-IFN 16 Weeks (Not Retreated): TDF 300 mg tablet once daily plus Peg-IFN 180 µg s.c. injection once weekly for 16 weeks followed by TDF 300 mg tablet once daily for an additional 32 weeks in the initial treatment phase
Arm/Group | TDF+Peg-IFN 48 Weeks (Not Retreated) | TDF+Peg-IFN 48 Weeks (Retreated) | TDF 48 Weeks + Peg-IFN 16 Weeks (Not Retreated) | TDF 48 Weeks + Peg-IFN 16 Weeks (Retreated) | TDF 120 Weeks | Peg-IFN 48 Weeks (Not Retreated) | Peg-IFN 48 Weeks (Retreated)
Number analyzed (Participants) | 144 | 42 | 131 | 53 | 185 | 128 | 57
percentage of participants | 15.3 | 26.2 | 14.5 | 15.1 | 84.9 | 11.7 | 40.4

9. Secondary Outcome: Percentage of Participants With Virological Response (HBV DNA < 117 IU/mL) at Week 96
Description: For the TDF+Peg-IFN 48 Weeks, TDF 48 Weeks + Peg-IFN 16 Weeks, and Peg-IFN 48 Weeks groups, data are presented in the "Not Retreated" column for participants who had not entered the retreatment phase by Week 96, and in the "Retreated" column for participants who did enter the retreatment phase by Week 96.
Time Frame: Week 96
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | TDF+Peg-IFN 48 Weeks (Not Retreated) | TDF+Peg-IFN 48 Weeks (Retreated) | TDF 48 Weeks + Peg-IFN 16 Weeks (Not Retreated) | TDF 48 Weeks + Peg-IFN 16 Weeks (Retreated) | TDF 120 Weeks | Peg-IFN 48 Weeks (Not Retreated) | Peg-IFN 48 Weeks (Retreated)
Number analyzed (Participants) | 83 | 103 | 83 | 101 | 185 | 72 | 113
percentage of participants | 21.7 | 68.0 | 15.7 | 80.2 | 83.8 | 13.9 | 70.8

10. Secondary Outcome: Percentage of Participants With Virological Response (HBV DNA < 117 IU/mL) at Week 120
Description: For the TDF+Peg-IFN 48 Weeks, TDF 48 Weeks + Peg-IFN 16 Weeks, and Peg-IFN 48 Weeks groups, data are presented in the "Not Retreated" column for participants who had not entered the retreatment phase by Week 120, and in the "Retreated" column for participants who did enter the retreatment phase by Week 120.
Time Frame: Week 120
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | TDF+Peg-IFN 48 Weeks (Not Retreated) | TDF+Peg-IFN 48 Weeks (Retreated) | TDF 48 Weeks + Peg-IFN 16 Weeks (Not Retreated) | TDF 48 Weeks + Peg-IFN 16 Weeks (Retreated) | TDF 120 Weeks | Peg-IFN 48 Weeks (Not Retreated) | Peg-IFN 48 Weeks (Retreated)
Number analyzed (Participants) | 74 | 112 | 69 | 115 | 185 | 68 | 117
percentage of participants | 32.4 | 81.3 | 18.8 | 83.5 | 82.2 | 13.2 | 82.1

11. Secondary Outcome: Percentage of Participants With Normal ALT at Week 72
Description: Normal ALT was ≤ 30 U/L for males and ≤ 19 U/L for females (based on the American Association for the Study of Liver Diseases (AASLD) 2008 guidelines), and ≤ 41 U/L for males and ≤ 31 U/L for females (based on central laboratory upper limit of the normal range (ULN) for ALT).
  For the TDF+Peg-IFN 48 Weeks, TDF 48 Weeks + Peg-IFN 16 Weeks, and Peg-IFN 48 Weeks groups, data are presented in the "Not Retreated" column for participants who had not entered the retreatment phase by Week 72, and in the "Retreated" column for participants who did enter the retreatment phase by Week 72.
Time Frame: Week 72
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Groups:
- Peg-IFN 48 Week (Not Retreated): Peg-IFN 180 µg s.c. injection once weekly for 48 weeks in the initial treatment phase
Arm/Group | TDF+Peg-IFN 48 Weeks (Not Retreated) | TDF+Peg-IFN 48 Weeks (Retreated) | TDF 48 Weeks + Peg-IFN 16 Weeks (Not Retreated) | TDF 48 Weeks + Peg-IFN 16 Weeks (Retreated) | TDF 120 Weeks | Peg-IFN 48 Week (Not Retreated) | Peg-IFN 48 Weeks (Retreated)
Number analyzed (Participants) | 126 | 60 | 118 | 66 | 185 | 120 | 65
percentage of participants
  AASLD Criteria | 42.1 | 18.3 | 40.7 | 18.2 | 47.6 | 35.0 | 9.2
  Central Laboratory Criteria | 59.5 | 40.0 | 57.6 | 34.8 | 72.4 | 57.5 | 33.8

12. Secondary Outcome: Percentage of Participants With Normal ALT at Week 96
Description: Normal ALT was ≤ 30 U/L for males and ≤ 19 U/L for females (based on the American Association for the Study of Liver Diseases (AASLD) 2008 guidelines), and ≤ 41 U/L for males and ≤ 31 U/L for females (based on central laboratory upper limit of the normal range (ULN) for ALT).
  For the TDF+Peg-IFN 48 Weeks, TDF 48 Weeks + Peg-IFN 16 Weeks, and Peg-IFN 48 Weeks groups, data are presented in the "Not Retreated" column for participants who had not entered the retreatment phase by Week 96, and in the "Retreated" column for participants who did enter the retreatment phase by Week 96.
Time Frame: Week 96
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | TDF+Peg-IFN 48 Weeks (Not Retreated) | TDF+Peg-IFN 48 Weeks (Retreated) | TDF 48 Weeks + Peg-IFN 16 Weeks (Not Retreated) | TDF 48 Weeks + Peg-IFN 16 Weeks (Retreated) | TDF 120 Weeks | Peg-IFN 48 Week (Not Retreated) | Peg-IFN 48 Weeks (Retreated)
Number analyzed (Participants) | 81 | 105 | 82 | 102 | 185 | 72 | 113
percentage of participants
  AASLD Criteria | 43.2 | 42.9 | 34.1 | 46.1 | 48.1 | 34.7 | 39.8
  Central Laboratory Criteria | 55.6 | 71.4 | 52.4 | 73.5 | 73.0 | 47.2 | 68.1

13. Secondary Outcome: Percentage of Participants With Normal ALT at Week 120
Description: Normal ALT was ≤ 30 U/L for males and ≤ 19 U/L for females (based on the American Association for the Study of Liver Diseases (AASLD) 2008 guidelines), and ≤ 41 U/L for males and ≤ 31 U/L for females (based on central laboratory upper limit of the normal range (ULN) for ALT).
  For the TDF+Peg-IFN 48 Weeks, TDF 48 Weeks + Peg-IFN 16 Weeks, and Peg-IFN 48 Weeks groups, data are presented in the "Not Retreated" column for participants who had not entered the retreatment phase by Week 120, and in the "Retreated" column for participants who did enter the retreatment phase by Week 120.
Time Frame: Week 120
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | TDF+Peg-IFN 48 Weeks (Not Retreated) | TDF+Peg-IFN 48 Weeks (Retreated) | TDF 48 Weeks + Peg-IFN 16 Weeks (Not Retreated) | TDF 48 Weeks + Peg-IFN 16 Weeks (Retreated) | TDF 120 Weeks | Peg-IFN 48 Week (Not Retreated) | Peg-IFN 48 Weeks (Retreated)
Number analyzed (Participants) | 74 | 112 | 69 | 115 | 185 | 68 | 117
percentage of participants
  AASLD Criteria | 39.2 | 54.5 | 30.4 | 48.7 | 48.6 | 30.9 | 47.0
  Central Laboratory Criteria | 44.6 | 72.3 | 40.6 | 78.3 | 73.0 | 41.2 | 73.5

14. Secondary Outcome: Percentage of Participants Who Required Retreatment
Description: Participants in the TDF 120 week group were not eligible to enter the retreatment phase and are not presented.
Time Frame: Up to 120 weeks
Population: Safety Analysis Set. Participants in the TDF+Peg-IFN 48 Weeks, TDF 48 Weeks + Peg-IFN 16 Weeks, and Peg-IFN 48 Weeks groups were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TDF+Peg-IFN 48 Weeks | TDF 48 Weeks + Peg-IFN 16 Weeks | Peg-IFN 48 Weeks
Number analyzed (Participants) | 186 | 184 | 185
percentage of participants | 60.2 | 62.5 | 63.2

ADVERSE EVENTS:
Time Frame: Up to 120 weeks plus 30 days
Description: Safety Analysis Set: participants who were randomized and received at least 1 dose of study drug. Participants were analyzed by actual treatment received.
Groups:
- TDF+Peg-IFN 48 Weeks (Not Retreated): Adverse events in this reporting group are those occurring in participants who were not retreated or before retreatment through last non-retreatment dose plus 30 days.
  TDF 300 mg tablet once daily plus Peg-IFN 180 µg s.c. injection once weekly for 48 weeks
- TDF+Peg-IFN 48 Weeks (Retreated); TDF 48 Weeks + Peg-IFN 16 Weeks (Retreated): Adverse events in this reporting group are those occurring after TDF retreatment through last TDF retreatment dose plus 30 days.
  TDF 300 mg tablet once daily up to Week 120
- TDF 48 Week + Peg-IFN 16 Weeks (Not Retreated): Adverse events in this reporting group are those occurring in participants who were not retreated or before retreatment through last non-retreatment dose plus 30 days.
  TDF 300 mg tablet once daily plus Peg-IFN 180 µg s.c. injection once weekly for 16 weeks followed by TDF 300 mg tablet once daily for an additional 32 weeks
- TDF 120 Weeks: Adverse events in this reporting group are those occurring during the initial treatment phase (up to 120 weeks plus 30 days).
  TDF 300 mg tablet once daily for up to 120 weeks
- Peg-IFN 48 Weeks (Not Retreated): Adverse events in this reporting group are those occurring in participants who were not retreated or before retreatment through last non-retreatment dose plus 30 days.
  Peg-IFN 180 µg s.c. injection once weekly for 48 weeks
- Peg-IFN 48 Weeks (Retreated): Adverse events in this reporting group are those occurring during the retreatment phase (from start of retreatment up to Week 120 plus 30 days).
  TDF 300 mg tablet once daily up to Week 120
Arm/Group | TDF+Peg-IFN 48 Weeks (Not Retreated) | TDF+Peg-IFN 48 Weeks (Retreated) | TDF 48 Week + Peg-IFN 16 Weeks (Not Retreated) | TDF 48 Weeks + Peg-IFN 16 Weeks (Retreated) | TDF 120 Weeks | Peg-IFN 48 Weeks (Not Retreated) | Peg-IFN 48 Weeks (Retreated)
Serious Adverse Events (participants affected / at risk) | 21/186 | 7/112 | 18/184 | 3/115 | 13/185 | 18/185 | 6/117
Other Adverse Events (participants affected / at risk) | 147/186 | 26/112 | 142/184 | 31/115 | 89/185 | 152/185 | 33/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TDF+Peg-IFN 48 Weeks (Not Retreated) (N=186) | TDF+Peg-IFN 48 Weeks (Retreated) (N=112) | TDF 48 Week + Peg-IFN 16 Weeks (Not Retreated) (N=184) | TDF 48 Weeks + Peg-IFN 16 Weeks (Retreated) (N=115) | TDF 120 Weeks (N=185) | Peg-IFN 48 Weeks (Not Retreated) (N=185) | Peg-IFN 48 Weeks (Retreated) (N=117)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial septal defect acquired (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 3 | 2 | 4 | 0 | 1 | 7 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Psoas abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 6 | 3 | 8 | 2 | 1 | 7 | 2
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 1 | 0 | 0 | 2 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cholesterosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gallbladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mixed hepatocellular cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myelopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TDF+Peg-IFN 48 Weeks (Not Retreated) (N=186) | TDF+Peg-IFN 48 Weeks (Retreated) (N=112) | TDF 48 Week + Peg-IFN 16 Weeks (Not Retreated) (N=184) | TDF 48 Weeks + Peg-IFN 16 Weeks (Retreated) (N=115) | TDF 120 Weeks (N=185) | Peg-IFN 48 Weeks (Not Retreated) (N=185) | Peg-IFN 48 Weeks (Retreated) (N=117)
Neutropenia (Blood and lymphatic system disorders) | 15 | 0 | 11 | 1 | 0 | 15 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 1 | 6 | 1 | 6 | 10 | 1
Abdominal pain upper (Gastrointestinal disorders) | 11 | 2 | 7 | 0 | 7 | 6 | 6
Diarrhoea (Gastrointestinal disorders) | 13 | 2 | 10 | 0 | 11 | 19 | 4
Dyspepsia (Gastrointestinal disorders) | 9 | 1 | 6 | 1 | 15 | 9 | 1
Nausea (Gastrointestinal disorders) | 26 | 0 | 24 | 3 | 11 | 13 | 6
Asthenia (General disorders) | 20 | 0 | 9 | 1 | 4 | 12 | 1
Chills (General disorders) | 5 | 0 | 13 | 0 | 3 | 11 | 1
Fatigue (General disorders) | 40 | 2 | 33 | 4 | 21 | 41 | 6
Influenza like illness (General disorders) | 19 | 0 | 17 | 0 | 10 | 17 | 2
Injection site erythema (General disorders) | 12 | 0 | 11 | 0 | 0 | 10 | 0
Malaise (General disorders) | 20 | 0 | 12 | 1 | 2 | 7 | 3
Pain (General disorders) | 8 | 0 | 5 | 0 | 0 | 11 | 2
Pyrexia (General disorders) | 39 | 1 | 36 | 1 | 8 | 43 | 2
Nasopharyngitis (Infections and infestations) | 5 | 3 | 16 | 3 | 20 | 6 | 3
Upper respiratory tract infection (Infections and infestations) | 10 | 3 | 9 | 9 | 16 | 10 | 5
Decreased appetite (Metabolism and nutrition disorders) | 23 | 0 | 36 | 2 | 2 | 18 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 3 | 11 | 3 | 4 | 9 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 3 | 11 | 3 | 11 | 10 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 2 | 1 | 10 | 8 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 29 | 0 | 36 | 1 | 2 | 35 | 1
Dizziness (Nervous system disorders) | 20 | 0 | 18 | 1 | 9 | 17 | 4
Headache (Nervous system disorders) | 54 | 3 | 37 | 3 | 16 | 52 | 4
Insomnia (Psychiatric disorders) | 19 | 3 | 14 | 1 | 6 | 18 | 2
Irritability (Psychiatric disorders) | 11 | 1 | 2 | 0 | 0 | 11 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 3 | 9 | 3 | 12 | 16 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 3 | 5 | 0 | 9 | 11 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 46 | 0 | 32 | 1 | 2 | 45 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 0 | 14 | 2 | 4 | 21 | 0
Rash (Skin and subcutaneous tissue disorders) | 20 | 1 | 17 | 1 | 1 | 9 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years